CLINICAL TRIAL: NCT04467957
Title: Non-contrast Lung Perfusion Mapping Applied for New Insights in Cystic Fibrosis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-1192
Record Dates: First submitted 2020-06-19; First posted 2020-07-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Cystic fibrosis transmembrane conductance regulator modulator therapy; hyperpolarized xenon; Cystic fibrosis transmembrane conductance regulator (CFTR)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CF Cohort (Experimental): 16 Cystic Fibrosis Patients will undergo MRI imaging before and 6 months after initiation of triple-combination modulator therapy. Initiation of triple -combination modulator therapy will be determined by clinician and family prior to study enrollment. Hyperpolarized Xenon 129 will be administered through inhalation at two MRI imaging study visits.
  Interventions: Drug: Initiation of CFTR Modulator; Drug: Hyperpolarized Xenon 129
- Control Cohort (Experimental): 10 Healthy control study participants matched for age and gender will undergo one MRI imaging study visit. Hyperpolarized Xenon 129 will be administered through inhalation at one MRI imaging study visit.
  Interventions: Drug: Hyperpolarized Xenon 129

INTERVENTIONS:
Drug: Initiation of CFTR Modulator — Inhaled contrast for MRI occurring at each visit
  Other Names: 129Xe
  Arms: CF Cohort
Drug: Hyperpolarized Xenon 129 — Inhaled contrast for MRI occurring at each visit
  Other Names: 129Xe

SUMMARY:
Cystic fibrosis (CF) results in the thickening of mucus in the lungs and other organs due to dysfunction of a transmembrane conductance protein. This allows buildup of bacteria that results in inflammation, leading to tissue breakdown and loss of function. In the lungs, this process causes loss of air exchange structures progressing to diminished lung function. The exchange of oxygen in the lungs depends on both the integrity of air conduits and vasculature. Most clinical assessments, however, focus on ventilatory function, with the assumption that any vascular compromise is secondary. Nevertheless, there is evidence, some from the investigator's lab, to suggest that perfusion anomalies in the lung occur before signs of ventilatory dysfunction. Thus, the inflammatory processes of CF may impact pulmonary microvasculature specifically and concurrently or prior to damage to ventilatory structures. This study aims to apply a new MRI method to serially measure regional lung perfusion, without the use of contrast agent, in children with CF and to associate it with regional assessments of ventilation and to serum cytokines or proteomic markers of angiogenesis and inflammatory processes.

The investigator's lab has recently developed a noninvasive, non-contrast, method of labeling blood flowing into the lungs and generating a map of perfusion. The investigator aims to couple this technique to existing methods using hyperpolarized Xenon to map ventilation. The investigator will apply these methods over time in CF patients, monitoring the relationship between regional perfusion and ventilation defects.

This pilot work will provide the foundation for larger studies to establish the essential etiological role of perfusion deficits in CF.

DETAILED DESCRIPTION:
The Lung Perfusion in CF trial is a case-control observational study conducted at Cincinnati Children's Hospital.

Patients will be assessed before and approximately 6 months after the clinical initiation of triple-combination modulator therapy with the following imaging to demonstrate aim 1, that pulmonary perfusion is regionally altered in CF patients in association with the status and progression of lung ventilatory function: Ultra-short echo time (UTE) protocol to obtain structural lung imaging primarily for anatomic reference, Hyperpolarized Xenon gas inhalation protocol to measure regional lung ventilation and arterial spin labeling protocol to measure regional lung perfusion.

To demonstrate aim 2, that different profiles of serum proteomic markers related to angiogenesis and vascular remodeling, characterize states of pulmonary hyperfusion and hypoperfusion, blood sample data analysis from a separate study conducted at Cincinnati Children's Hospital Medical Center will also be obtained before and 6 months after initiation of triple-combination modulator therapy.

Safety will be assessed by recording adverse events. Vital signs (heart rate, SPO2) will be recorded before, immediately following inhalation, and 2 minutes after each Xenon gas inhalation; O2 saturation will be monitored continuously throughout the Xenon portion of the MRI, and the time and duration of nadir will be recorded.

The overarching goal of this study is to demonstrate that arterial spin labeling MRI lung perfusion can be used to measure regional manifestations of pulmonary vascular disease in CF that precedes and contributes to global and local decline in ventilatory lung function.

ELIGIBILITY:
Inclusion Criteria:

Inclusion CF Cohort

* male or female between the ages of 6 through 21 years
* diagnosis of CF by positive sweat test and genetic test
* planning to start Trikafta based on clinical decision
* baseline pulmonary function test (PFT) defined as FEV1% that is no less than 5% of the best PFT in the previous 6 months
* Absence of exacerbation defined as

  * No acute antibiotic usage for 14 days prior to MRI visit
  * Able to perform an acceptable and reproducible spirometry
  * O2 saturation level at 90% or greater when laying flat

Inclusion Healthy Control Cohort

* male or female between the ages of 6 through 21 years
* no known diagnoses that impact lung function in the opinion of the investigators

Exclusion Criteria:

Exclusion both cohorts

* standard MRI exclusions (metal implants, claustrophobia)
* pregnancy

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percentage (VDP) | Baseline and 6 months post Trikafta initiation for CF group. Baseline for CF and control groups.
  Lung defect calculations (total and lobar defect percentages) will be performed by evaluating the percentage of voxels with signals below a threshold value of 60% of the total lung mean signal. This threshold (60%) represents our estimate of the visually accurate defect selection threshold for CF patients. To assign the pixels in the hyperpolarized Xenon gas (129Xe) MRI slices to a lobe, corresponding CT and/or UTE MRI images will be segmented and analyzed with custom MATLAB software.
  VDP for CF and Control groups will be compared by 2-sample T-test at baseline. VDP at baseline and 6 months for the CF group will be compared by paired T-test to determine if the change is significantly different from zero change.
Perfusion Defect Percentage (PDP) | Baseline and 6 months post Trikafta initiation for CF group. Baseline for CF and control groups.
  Similar to the VDP, total and lobar defect percentages will be calculated for lung perfusion.
  As for VDP, PDP will be compared between CF and Control groups at baseline via 2-sample T-test.
  PDP change from baseline to 6 months will be measured for the CF group via paired T-test to determine change significantly different from zero change.
Degree of concordance between ventilation and perfusion defects | Baseline and 6 months post Trikafta initiation for CF group. Baseline for CF and control groups.
  Degree of concordance between ventilation and perfusion defects will be calculated as percentage of overlap between ventilation and perfusion defect volumes.
Proteome assays as global indicators of inflammatory/angiogenic processes | Baseline and 6 months post Trikafta initiation for CF group. Baseline for CF and control groups.
  Proteome assays as global indicators of inflammatory/angiogenic processes, will be compared between groups by 2-sample T-test. Correlation analyses will be performed to examine associations between quantitative image scores for each modality (VDP and PDP) and lung function (FEV1%), as well as proteome concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Mark DiFrancesco, PhD, Principal Investigator — CCHMC; Jason Woods, PhD, Study Chair — CCHMC
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No